CLINICAL TRIAL: NCT00435487
Title: Prospective Randomized Phase IV Open Label Comparative Study Of Dalteparin vs Unfractionated Heparin In High Risk Patients Of Non-ST Elevation Acute Coronary Syndromes Intended For Early Invasive Strategy
Brief Title: Dalteparin Versus Unfractionated Heparin In Patients With Acute Coronary Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6301079
Record Dates: First submitted 2007-02-13; First posted 2007-02-15 (Estimated); Results first posted 2010-01-27 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Angina, Unstable; Myocardial Infarction
Keywords: Non-ST Elevation Acute Coronary Syndromes coronary interventions
MeSH Terms: conditions — Angina, Unstable; Myocardial Infarction | interventions — Dalteparin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Dalteparin ( Fragmin)
- B (Active Comparator)
  Interventions: Drug: Unfractionated heparin

INTERVENTIONS:
Drug: Dalteparin ( Fragmin) — Dalteparin will be administered at a dose of 120 IU/kg (international units per kilogram) total body weight subcutaneously (SC) every 12 hours up to a maximum dose of 10,000 IU/12 hours.
  Arms: A
Drug: Unfractionated heparin — Unfractionated heparin will be given intravenously according to a weight-adjusted nomogram (bolus of 60 U/kg [units per kilogram] and initial infusion of 12 U/kg/h [units per kilogram per hour]).
  Arms: B

SUMMARY:
To compare efficacy and safety of dalteparin compared to unfractionated heparin in patients of non ST elevation acute coronary syndromes who are planned to undergo coronary interventions (angioplasty or bypass surgery)

DETAILED DESCRIPTION:
The study was prematurely discontinued on November 30, 2008 due to delay in meeting pre-defined protocol recruitment milestones. There were no safety concerns regarding the study in the decision to terminate the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years
* Ischemic pain of more than 10 minutes within 24 hours before enrollment
* At least two of the following three risk factors : Age more than 60 years ( or more than 50 in case of diabetics), Raised cardiac enzyme levels, abnormal ECG findings

Exclusion Criteria:

* Contraindications to use of anticoagulants
* Active bleeding or abnormal coagulation tests
* Ischemic stroke within last 6 months or hemorrhagic stroke
* Lumbar or spinal puncture within last 48 hours
* S creatinine levels more than 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- India (6):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Nagpur, Maharashtra
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Ludhiana, Punjab
  - Pfizer Investigational Site, Coimbatore, Tamil Nadu
  - Pfizer Investigational Site, Karnataka

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6301079&StudyName=Dalteparin%20Versus%20Unfractionated%20Heparin%20In%20Patients%20With%20Acute%20Coronary%20Syndrome

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects participated in the study between 22 June 2007 and 30 December 2008.
Groups:
- Arm A: Dalteparin: 120 international units per kilogram (IU/kg) total body weight subcutaneously (SC) every 12 hours up to a maximum dose of 10,000 IU/12 hours; given for a minimum of 48 hours and until no further anticoagulation is required, and at least through angiography and percutaneous coronary intervention (PCI), if performed.
- Arm B: Unfractioned Heparin (UFH): Weight-adjusted nomogram (bolus of 60 units per kilogram [U/kg] and initial infusion of 12 units per kilogram per hour [U/kg/h]); given for a minimum of 48 hours and until no further anticoagulation is required, and at least through angiography and percutaneous coronary intervention (PCI), if performed.
Period: Overall Study
Arm/Group | Arm A: Dalteparin | Arm B: Unfractioned Heparin (UFH)
Started | 88 (87 subjects were randomized however one additional subject originally randomized to UFH was treated.) | 86
TREATED | 88 (One additional subject originally randomized to Unfractioned Heparin was treated with Dalteparin.) | 83 (One subject was mistakenly treated with Dalteparin, two subjects withdrew consent before treatment.)
Completed | 76 | 71
Not Completed | 12 | 15
Not completed — Death | 3 | 4
Not completed — Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Other | 5 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Withdrawal by Subject Prior to Treatment | 0 | 2
Not completed — Received Drug in Other Treatment Group | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Dalteparin | Arm B: Unfractioned Heparin (UFH) | Total
Number analyzed (Participants) | 88 | 83 | 171
Age, Customized [Number; unit: participants]
  18 - 44 years | 6 | 5 | 11
  45 - 64 years | 36 | 40 | 76
  >=65 years | 46 | 38 | 84
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 40 | 69
  Male | 59 | 43 | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Death or Non-fatal Myocardial Infarction Through and Up to Day 30
Description: Death or non-fatal myocardial infarction (MI) after receiving 48 hours of study medication (event date - first dose date) on or before day 30 from baseline. Death: fatal event resulting from any cause. New MI: electrocardiographic (ECG) and or biomarker criteria of myocardial necrosis. Biochemical markers: creatine phosphokinase - myocardial band (CPK-MB) levels and the qualitative troponin-T test.
Time Frame: Baseline to Day 30
Population: Evaluable population: all subjects who took study medication for at least 48 hours from baseline and had complete information on the endpoint.
Measure: Number; unit: participants
Arm/Group | Arm A: Dalteparin | Arm B: Unfractioned Heparin (UFH)
Number analyzed (Participants) | 79 | 78
participants
  Death | 2 | 4
  Non-fatal Myocardial Infarction | 2 | 1
  Death or Non-fatal Myocardial Infarction | 4 | 5
Statistical Analysis 1: Comparison: Arm A: Dalteparin vs Arm B: Unfractioned Heparin (UFH); Death after receiving 48 hours of study medication (Event date - First dose date) and on or before day 30 from baseline. Difference in proportion (Dalteparin-UFH)(%); Test type: Non-Inferiority or Equivalence — The test of non-inferiority was based on whether the upper limit of the two-sided 95% confidence interval for the treatment group difference was less than or equal to 10%, the non-inferiority margin specified in the protocol; upper limit of 95% CI <= 10%; Difference in proportion = -2.60, 95% CI [-8.59 to 3.40] — 95% confidence interval (CI) is for difference in proportion using normal approximation to binomial. Non-inferiority was concluded if the upper boundary of the 95% CI for the Dalteparin - Unfractioned Heparin difference was less than or equal to 10%
Statistical Analysis 2: Comparison: Arm A: Dalteparin vs Arm B: Unfractioned Heparin (UFH); Non-fatal Myocardial Infarction after receiving 48 hours of study medication (Event date - First dose date) and on or before day 30 from baseline. Difference in proportion (Dalteparin-UFH)(%); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; upper limit of 95% CI <= 10%; Difference in proportion = 1.25, 95% CI [-3.02 to 5.52] — 95% CI is for difference in proportion using normal approximation to binomial. Non-inferiority was concluded if the upper boundary of the 95% CI for the Dalteparin - Unfractioned Heparin difference was less than or equal to 10%
Statistical Analysis 3: Comparison: Arm A: Dalteparin vs Arm B: Unfractioned Heparin (UFH); Death or Non-fatal Myocardial Infarction after receiving 48 hours of study medication (Event date - First dose date) and on or before day 30 from baseline. Difference in proportion (Dalteparin-UFH)(%); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; upper limit of 95% CI <= 10%; Difference in proportion = -1.35, 95% CI [-8.62 to 5.93] — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Number of Subjects With Stroke
Description: Stroke: a sudden, focal neurologic deficit that is not reversible within 24 hours and is not the result of any readily identifiable cause (e.g., tumor or trauma).
Time Frame: End of hospitalization, Day 30
Population: Evaluable population
Measure: Number; unit: participants
Arm/Group | Arm A: Dalteparin | Arm B: Unfractioned Heparin (UFH)
Number analyzed (Participants) | 79 | 78
participants | 1 | 0
Statistical Analysis 1: Comparison: Arm A: Dalteparin vs Arm B: Unfractioned Heparin (UFH); Difference in proportion (Dalteparin-UFH)(%); Test type: Superiority or Other; p = 1.0000, Chi-squared; Difference in proportion = 1.27, 95% CI [-1.20 to 3.73] — 95% CI is for difference in proportion using normal approximation to binomial

3. Secondary Outcome: Number of Subjects With Recurrent Angina With or Without Need for Hospitalization and or Revascularization
Description: Recurrent angina: angina at rest lasting at least five minutes that was associated with a new ST-segment shift (elevation or depression) of more than 0.1 millivolt (mV), or with T-wave inversions, in two contiguous electrocardiographic leads; angina without electrocardiographic changes that prompted a decision to perform a revascularization procedure; or angina after hospital discharge that resulted in rehospitalization.
Time Frame: End of hospitalization, Day 30
Population: Evaluable population
Measure: Number; unit: participants
Arm/Group | Arm A: Dalteparin | Arm B: Unfractioned Heparin (UFH)
Number analyzed (Participants) | 79 | 78
participants | 3 | 3
Statistical Analysis 1: Comparison: Arm A: Dalteparin vs Arm B: Unfractioned Heparin (UFH); Difference in proportion (Dalteparin-UFH)(%); Test type: Superiority or Other; p = 1.0000, Chi-squared; Difference in proportion = -0.05, 95% CI [-6.05 to 5.95] — 95% CI is for difference in proportion using normal approximation to binomial

4. Secondary Outcome: Number of Subjects With Death or Non-fatal Myocardial Infarction (MI), Computed Separately, at End of Hospitalization and 30 Days
Description: Death or non-fatal myocardial infarction (MI) after receiving 48 hours of study medication (event date - first dose date) at end of hospitalization and on Day 30. Death: fatal event resulting from any cause. New MI: defined by electrocardiographic and/or biomarker criteria of myocardial necrosis. Biochemical markers: creatine phosphokinase - myocardial band (CPK-MB) levels and the qualitative troponin-T test.
Time Frame: End of hospitalization, Day 30
Population: Evaluable population
Measure: Number; unit: participants
Arm/Group | Arm A: Dalteparin | Arm B: Unfractioned Heparin (UFH)
Number analyzed (Participants) | 79 | 78
participants | 3 | 3
Statistical Analysis 1: Comparison: Arm A: Dalteparin vs Arm B: Unfractioned Heparin (UFH); Difference in proportion (Dalteparin-UFH)(%); Test type: Superiority or Other; p = 1.0000, Chi-squared; Difference in proportion = -0.05, 95% CI [-6.05 to 5.95] — 95% CI is for difference in proportion using normal approximation to binomial

5. Secondary Outcome: Number of Subjects With Stent Thrombosis and Abrupt Closures During Hospitalization
Description: Abrupt vessel closure and or stent thrombosis: occurrence of vessel closure (no visible antegrade flow of contrast dye occurring after balloon angioplasty) or stent thrombosis determined angiographically.
Time Frame: End of hospitalization, Day 30
Population: Evaluable population
Measure: Number; unit: participants
Arm/Group | Arm A: Dalteparin | Arm B: Unfractioned Heparin (UFH)
Number analyzed (Participants) | 79 | 78
participants | 0 | 0

6. Secondary Outcome: Number of Subjects With Bleeding by Thrombolysis in Myocardial Infarction (TIMI) Criteria
Description: Thrombolysis in myocardial infarction (TIMI) major bleeding: at least a 5-grams per deciliter (g/dL) decrease in hemoglobin, at least a 15 percent (%) decrease in hematocrit, or intracranial bleeding. TIMI minor bleeding: associated with gastrointestinal or genitourinary bleeding, with an absolute decrease in hemoglobin of 4 g/dL or more, or decrease in hematocrit of at least 12%.
Time Frame: End of hospitalization, Day 30
Population: Evaluable population
Measure: Number; unit: participants
Arm/Group | Arm A: Dalteparin | Arm B: Unfractioned Heparin (UFH)
Number analyzed (Participants) | 79 | 78
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm A: Dalteparin | Arm B: Unfractioned Heparin (UFH)
Serious Adverse Events (participants affected / at risk) | 4/88 | 13/83
Other Adverse Events (participants affected / at risk) | 58/88 | 59/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Dalteparin (N=88) | Arm B: Unfractioned Heparin (UFH) (N=83)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 2
Collapse of lung (Injury, poisoning and procedural complications) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Dalteparin (N=88) | Arm B: Unfractioned Heparin (UFH) (N=83)
Anaemia (Blood and lymphatic system disorders) | 4 | 5
Angina pectoris (Cardiac disorders) | 4 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac asthma (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 3
Palpitations (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Eye pain (Eye disorders) | 0 | 1
Pseudophakia (Eye disorders) | 0 | 1
Retinopathy hypertensive (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 9
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 6
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 4
Asthenia (General disorders) | 1 | 2
Chest pain (General disorders) | 9 | 6
Chills (General disorders) | 1 | 1
Facial pain (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 4
Pain (General disorders) | 3 | 0
Puncture site reaction (General disorders) | 0 | 1
Pyrexia (General disorders) | 13 | 9
Pneumonia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 3
Blood creatinine increased (Investigations) | 2 | 1
Blood pressure increased (Investigations) | 1 | 0
ECG signs of myocardial ischaemia (Investigations) | 0 | 2
Electrocardiogram ST segment depression (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Venous pressure jugular increased (Investigations) | 2 | 2
White blood cell count increased (Investigations) | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Joint crepitation (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 4 | 10
Syncope (Nervous system disorders) | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 4 | 4
Insomnia (Psychiatric disorders) | 1 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 2
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal disorder (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 1
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 3
Ischaemia (Vascular disorders) | 0 | 2
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated due to insufficient recruitment of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.